CLINICAL TRIAL: NCT03195868
Title: A Comparative Analysis of Changes in Peripheral Nerve Density and Structure Following Photobiomodulation Therapy Using the REALief Therapy System for Patients With Diabetic or Chemotherapy-associated Neuropathy
Brief Title: Photobiomodulation Therapy and Nerve Density for Patients With Diabetic or Chemotherapy-associated Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017NTLS037
Record Dates: First submitted 2017-06-01; First posted 2017-06-22 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Neuropathy; Neuropathy, Diabetic; Neuropathy Toxic
Keywords: chemotherapy; chemo-induced; CIPN
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: Single group, prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Photobiomodulation (Experimental): All patients will be treated similarly in this study
  Interventions: Device: Realief Therapy

INTERVENTIONS:
Device: Realief Therapy — Patients will be treated using class IV laser using a proprietary algorithm developed by REALief neuropathy centers
  Other Names: biopsies (skin, diagnostic not therapeutic)

SUMMARY:
This study seeks to determine if photobiomodulation (PBM, or low level laser light) affects the growth and distribution of nerves int he skin. Our previous study demonstrated that the treatment we use here was effective at reducing the symptoms of neuropathy (as measured by the modified total neuropathy score) in patients who had been treated with chemotherapy. The current effort is designed to repeat this confirm this observation using a more extensive battery of survey as well as to begin to elucidate the mechanism through which photobiomodulaiton produces the effect. WE will also be attempting to determine if diabetic patients differ in terms of response from chemotherapy patients

DETAILED DESCRIPTION:
Consenting patients with self-reported neuropathy following either diabetes or administration of chemotherapy, will undergo sensory testing and skin biopsies of the the foot and leg prior to initiating treatment. They will undergo PBM 3 times weekly for 6 weeks with with a follow-up biopsy performed at the conclusion of therapy and sensory testing throughout. Patients will have one remote evaluation at 26 weeks to determine whether the effect, if any extinguishes.

ELIGIBILITY:
Inclusion Criteria: self reported neuropathy following exposure to diabetes or chemotherapy

* willingness to undergo biopsies and 6 weeks of therapy

Exclusion Criteria:

* pregnancy
* active cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
change in epidermal nerve density and/or distribution | Change at Baseline 6 weeks, 26 weeks
  nerve measures include epidermal penetration points
total nerve fiber density, | Change at Baseline 6 weeks, 26 weeks
  nerve measures

SECONDARY OUTCOMES:
Brief Pain index | Change at Baseline 6 weeks, 26 weeks
NTSS- Nueropathy Total Symptom Score | Change at Baseline 6 weeks, 26 weeks
  This is a 15 question survey with yes or no answers. Averaged for scoring

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Argenta PA, Ballman KV, Geller MA, Carson LF, Ghebre R, Mullany SA, Teoh DG, Winterhoff BJ, Rivard CL, Erickson BK. The effect of photobiomodulation on chemotherapy-induced peripheral neuropathy: A randomized, sham-controlled clinical trial. Gynecol Oncol. 2017 Jan;144(1):159-166. doi: 10.1016/j.ygyno.2016.11.013. Epub 2016 Nov 22. PMID 27887804